CLINICAL TRIAL: NCT04362644
Title: Molecular Imaging Probes to Inform Heterogeneity in Idiopathic Pulmonary Fibrosis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Jonathan E McConathy, M.D. P.h.D., Director for the Division Molecular Imaging and Therapeutics, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: R20-010; 3109239 (Other Grant/Funding Number: UAB Pulmonology)
Record Dates: First submitted 2020-03-02; First posted 2020-04-27 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- PET/CT using PET ligands [18F]FDG and [18F]DPA-714 (Experimental)
  Interventions: Drug: PET/CT using PET ligands [F-18]FDG and [F-18]DPA-714

INTERVENTIONS:
Drug: PET/CT using PET ligands [F-18]FDG and [F-18]DPA-714 — Study participants will undergo PET/CT with the glucose analogue [F-18]FDG and the translocator protein (TSPO) ligand [F-18]DPA-714 in two separate imaging sessions.

SUMMARY:
The purpose of the study is to see if imaging with fluorine-18 Fluorodeoxyglucose ([18F] FDG) and fluorine-18 Displacement Per Atom ([18F]DPA-714) using positron emission tomography and computed tomography (PET/CT) will show lung inflammation and fibrosis in patients diagnosed with idiopathic pulmonary fibrosis (IPF). This study may help physicians and researchers better understand how best to treat patients with IPF in the future.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 40-85 years old.
2. A diagnosis of IPF that fulfills American Thoracic Society (ATS) / European Respiratory Society (ERS) 2018 consensus criteria within 5 years.
3. Ability and willingness to give informed consent and adhere to study requirements.
4. Ratio of forced expiratory volume in 1 second to forced vital capacity (FEV1/FVC) >0.70.
5. High or mixed affinity binder for TSPO ligands based on genotyping for single-nucleotide polymorphism (SNP)rs6971.

Exclusion Criteria:

1. Acute exacerbation of IPF within <30 days
2. Diagnosis of Diabetes Mellitus (Type 1 or Type 2).
3. Diagnoses of current infection by clinical or microbial assessments.
4. Treatment for >14 days within the preceding month with >20 mg. prednisone (or equivalent) or any treatment during the last month with a cellular immunosuppressant.
5. Subjects with prior radiation therapy to the thorax.
6. Women who are pregnant, or who are breastfeeding. IPF is a disease of older adults, and male predominant, so this will not be a frequent consideration.
7. Severe cardiovascular disease, defined as any of the following within the preceding 12 weeks: acute myocardial infarction or unstable angina, a coronary revascularization procedure, or stroke.
8. Subjects with known liver disease.
9. Diagnosis of any active cancer with the exception of basal cell carcinoma of skin.
10. Low affinity binder for TSPO ligands based on genotyping for SNP rs6971.
11. Active cigarette smoking or vaping

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-12-08 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Correlate quantitative PET measures of lung inflammation with [F-18]FDG and [F-18]DPA-714 to pulmonary function tests. | screening to 48 hours post 2nd imaging visit.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No